CLINICAL TRIAL: NCT05243654
Title: Efficacy and Tolerability of Adjunct Metformin in Combination With Multidrug Treatment for Multibacillary Leprosy: A Randomized Double-blind, Controlled Proof-of-Concept Phase 2 Trial in Indonesia
Brief Title: Efficacy and Tolerability of Adjunct Metformin for Multibacillary Leprosy
Acronym: MetLep
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit Indonesia (Other)
Collaborators: University of Gadjah Mada, Faculty of Medicine (Unknown); University of Diponegoro (Unknown); Papua Agency of Health Research and Development (NIHRD) (Unknown); London School of Hygiene and Tropical Medicine (Other); Radboud University Medical Center (Other); Oxford University Clinical Research Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EOCRU.2021.002; OXTREC 14-21 (Other: Oxford Tropical Research Ethics Committee)
Record Dates: First submitted 2021-09-30; First posted 2022-02-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Leprosy; Leprosy, Multibacillary; Neglected Tropical Diseases
Keywords: Leprosy; Multibacillary leprosy; Skin-NTD
MeSH Terms: conditions — Leprosy; Leprosy, Multibacillary; Neglected Diseases | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized double-blind, controlled phase 2 proof-of-concept trial. Subjects will be randomised 1:1 ratio to receive metformin 1000 mg XR tablets OD or matching placebo for 24 weeks. Randomization will be stratified by BI (BI ≥ or < 4) and participating study site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain blinding to treatment allocation, all subjects will receive treatment with identical tablets and the same number of tablets (two tablets once daily).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin 1000mg extended release (XR) once daily + standard-of-care MDT (Experimental): Metformin hydrochloride 500mg XR tablets once daily by mouth for 2 weeks, escalating to a target dose of 1000mg XR once daily for another 22 weeks. Each participant will receive the same number of tablets made up of metformin and placebo to maintain the blinding.
  Interventions: Drug: Metformin
- Placebo + MDT (Placebo Comparator): Matching metformin placebo tablets once daily by mouth for 2 weeks, escalating to two tablets for another 22 weeks. Each participant will receive the same number of tablets made up of metformin and placebo to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg XR OD + standard-of-care MDT
  Other Names: Glumin XR
  Arms: Metformin 1000mg extended release (XR) once daily + standard-of-care MDT
Drug: Placebo — Placebo + standard-of-care MDT
  Arms: Placebo + MDT

SUMMARY:
This trial aims to evaluate the efficacy, tolerability and safety of adjunct metformin added to standard-of-care multi-drug therapy (MDT) in patients with multibacillary leprosy, and explore its effects on immunological endpoints. A double-blind, placebo controlled proof-of-concept trial will be performed in which patients with newly diagnosed multibacillary leprosy will be randomized (1:1) to metformin 1000mg OD versus placebo for 24 weeks in addition to MDT during 48 weeks.

The main research question is whether adjunctive metformin, combined with MDT, will improve the clinical outcomes of patients with multibacillary leprosy by mitigating leprosy reactions, thereby reducing nerve damage and corticosteroid use and its associated morbidity. The second aim is to explore whether adjunct metformin, added to MDT, has an acceptable tolerability and safety in patients with multibacillary leprosy.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled randomized proof-of-concept Phase 2 trial will be performed evaluating the efficacy, safety and tolerability of adjunct metformin combined with standard of care MDT to mitigate leprosy reactions. Patients with newly diagnosed multibacillary leprosy will be randomized (1:1) to metformin 1000mg OD versus placebo for 24 weeks in addition to MDT during 48 weeks. The trial aims to enroll 166 patients, aged between 18-65 years old, in leprosy endemic areas in Indonesia. Primary endpoints are the proportion of participants experiencing a leprosy reaction during the full duration of the study and the proportion of participants with at least one adverse event within the first 28 weeks of the study. Secondary endpoints are the severity and time to first leprosy reaction, the number of leprosy reactions, the cumulative corticosteroid usage, and quality of life. The total study follow-up is 48 weeks.

This METLEP trial is financially supported by the Leprosy Research Initiative (grant number: FP20\4).

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female, aged ≥18 and ≤65 years.
* Participant is newly diagnosed with MB leprosy and has been receiving MDT ≤ 28 days.
* Participant is willing and able to give informed consent for participation in the trial.
* Participant is willing to adhere to study follow-up schedule for 48 weeks.

Exclusion Criteria:

* Participant has received MDT >28 days for the current episode of MB leprosy, prior to study enrolment.
* Presence of leprosy reaction and/or nerve function impairment requiring systemic corticosteroids on screening/enrolment evaluation.
* Participants who have been treated for leprosy in the past.
* Chronic systemic corticosteroid use for any other medical condition on screening evaluation (chronic use defined as ≥ 2 weeks).
* History of diabetes mellitus or diabetes mellitus diagnosed on screening evaluation (random blood glucose is elevated ≥200 mg/dL (or ≥11,1 mmol/L) or fasting blood glucose ≥ 126 mg/dL (or ≥7.0 mmol/L)).
* History of hypoglycaemia (random blood glucose <55 mg/dL (or <3.0 mmol/L).
* History of cardiac failure, ischaemic heart disease, alcoholism, history of lactic acidosis or states associated with lactic acidosis such as shock or pulmonary insufficiency, and conditions associated with hypoxia.
* History of intolerance or hypersensitivity to metformin.
* Estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73m2 calculated by the CKDEPI equation.
* AST or ALT ≥3 times the upper limit of normal (ULN) on screening evaluation.
* Any serious medical condition for which participation in the trial, as judged by the investigator or treating physician, could compromise the well-being of the subject or prevent, limit or confound protocol-specified assessments.
* HIV-positive on screening evaluation.
* Female participant of childbearing age who is pregnant (clinically confirmed or urine dipstick for human chorionic gonadotrophin hormone) or breastfeeding.
* Use of metformin within 12 weeks prior to study enrolment.
* Use of other regular hypoglycaemic agents, including insulin.
* Participation in another research trial involving an investigational product within 12 weeks prior to study enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants experiencing a leprosy reaction | 48 weeks
  Proportion of participants experiencing a leprosy reaction during study follow-up
The proportion of participants with at least one adverse events | 28 weeks
  The proportion of participants with at least one adverse events within the first 28 weeks of the study

SECONDARY OUTCOMES:
The proportion of participants experiencing a Type 1 Reactions (T1R) | 12, 24 and 48 weeks
  Proportion of participants experiencing a T1R at 12, 24 and 48 weeks.
The proportion of participants experiencing a Type 2 Reactions (T2R) | 12, 24 and 48 weeks
  Proportion of participants experiencing a T2 R at 12, 24 and 48 weeks.
The time to the first leprosy reaction | 48 weeks
  Time to first leprosy reaction over the full 48 weeks.
The time to the first Type 1 Reactions (T1R) | 48 weeks
  Time to first T1R over the full 48 weeks.
The time to the first Tipe 2 Reaction (T2R) | 48 weeks
  Time to first T2R over the full 48 weeks.
The difference in the number of T1R episodes | 48 weeks
  The difference in the number of T1R episodes
The difference in the number of T2R episodes | 48 weeks
  The difference in the number of T2R episodes
The severity of T1R, based on investigator-assessed validated Clinical Severity Scores | 48 weeks
  The severity of T1R based on the Modified Type 1 Reactions Clinical Severity Scale. The score ranges from 0-48. A higher score means a worse outcome.
The severity of T2R, based on investigator-assessed validated Clinical Severity Scores | 48 weeks
  The severity of T2R based on the ENLIST ENL Severity Scale. The score ranges from 0-30. A higher score means a worse outcome.
The proportion of participants with at least one serious adverse event | 28 weeks
  The proportion of participants with at least one serious adverse event within the first 28 weeks of the trial.
Total number of adverse events | 28 weeks
  The total number of adverse events within the first 28 weeks of the trial.
The cumulative corticosteroid usage | 48 weeks
  Cumulative corticosteroid usage over the full 48 weeks.
The proportion of participants experiencing clinical nerve function impairment | 48 weeks
  Proportion of participants experiencing clinical nerve function impairment developed over the full duration of the study.
The difference in Quality of Life between start and end of treatment intervention, and end of study by means of SF-36 questionnaires | 24 and 48 weeks
  The difference in Quality of Life between start and end of treatment intervention, and end of study by means of the 36-Item short form survey instrument (SF-36). This is a 36-item patient-reported questionnaire that covers eight health domains. Scores for each domain are 0 to 100, with a higher score defining a more favorable health state (0 points means maximum impact on quality of life, 100 means no impact on quality of life).
The difference in Quality of Life between start and end of treatment intervention, and end of study by means of the Dermatology Life Quality Index (DLQI) questionnaires. | 24 and 48 weeks
  The difference in Quality of Life between start and end of treatment intervention, and end of study by means of the Dermatology Life Quality Index (DLQI).
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0 points. A higher score defines a less favorable health state and the more quality of life is impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Hardiyanto Soebono, Prof.Dr.dr, Principal Investigator — Center of Tropical Medicine, University of Gadjah Mada
Locations (6):
- Indonesia (6):
  - Sitanala Leprosy Hospital, Tangerang, Banten
  - Palangga Health Center, Makassar, South Sulawesi
  - Bajeng Health Center, Makassar, South Sulawesi
  - Abe Pantai Community Health Center, Jayapura, Special Region of Papua
  - Hamadi Community Health Center, Jayapura, Special Region of Papua
  - Jayapura Utara Community Health Center, Jayapura, Special Region of Papua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krismawati H, Muchtar SV, Rahardjani M, Utami NN, Oktaviani M, Puspatriani K, Syamsiah, Imbiri N, Hasvitasari DE, Fajrianti DR, Tarino N, Wulandari F, Kestelyn E, Du DH, van Crevel R, Walker SL, Geskus RB, Geluk A, Hamers RL, Soebono H, Grijsen ML. Metformin as adjunctive therapy in combination with multidrug treatment for multibacillary leprosy: A protocol for a randomized double-blind, controlled Phase 2 trial in Indonesia (MetLep Trial). Wellcome Open Res. 2024 May 9;8:289. doi: 10.12688/wellcomeopenres.19455.2. eCollection 2023. PMID 38808319